CLINICAL TRIAL: NCT03259841
Title: Ultrasound Assessment of Gastric Contents in Fasted Patient Undergoing Cholecystectomy
Status: Completed | Type: Observational
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, associate professor, SMG-SNU Boramae Medical Center
Other Study IDs: 2017-8-4
Record Dates: First submitted 2017-08-04; First posted 2017-08-24 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fasted patients for cholecyctectomy: The fasted patients for cholecyctectomy except exclusion criteria are included
  Interventions: Other: Ultrasound assessment of gastric contet

INTERVENTIONS:
Other: Ultrasound assessment of gastric contet — Ultrasound assessment of gastric content is performed in fasted patient undergoing cholecystectomy.

SUMMARY:
Investigators assess the gastric contents by ultrasonography in fasted patients undergoing cholecystectomy.

DETAILED DESCRIPTION:
Investigators evaluate the gastric volume through cross sectional area and amount of clear fluid using Perlas grade by ultrasound in the supine and right lateral position of fasted patients undergoing cholecystectomy. Full stomach is regarded if solid gastric contents are detected or clear fluid is more than 1.5 ml/kg. The frequency of full stomach will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for cholecystectomy

Exclusion Criteria:

* Presence of gastric anatomic abnormality or pathology
* A previous surgery of esophagus or stomach
* Current pregnancy
* Who could not lie in the right lateral decubitus (RLD) position

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for cholecystectomy are included.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2019-02-08 (Actual)

PRIMARY OUTCOMES:
Incidence of full stomach | Before the induction of anesthesia
  The incidence of full stomach is assessed by using ultrasonography.

SECONDARY OUTCOMES:
Cross sectional area of the stomach | Before the induction of anesthesia
  The cross sectional area of the stomach is assessed by using ultrasonography in the supine and right lateral positions.
Volume of stomach | Before the induction of anesthesia
  The volume of stomach is assessed using the following formula; volume of stomach (mL) = 27.0 + 14.6 x cross-sectional area (right lateral position) - 1.28 x age.
Type of gastric contents | Before the induction of anesthesia
  The type of gastric contents is assessed using ultrasonography.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Young Hwang, M.D., Ph.D., Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang JE, Kim H, Won D, Lee JM, Jung JY, Min SW, Hwang JY. Ultrasound assessment of gastric content in fasted patients before elective laparoscopic cholecystectomy: a prospective observational single-cohort study. Can J Anaesth. 2020 Jul;67(7):810-816. doi: 10.1007/s12630-020-01668-7. Epub 2020 Apr 20. PMID 32314262